CLINICAL TRIAL: NCT06967935
Title: Rehearsal-Induced Memory Consolidation and Its Modulation by Sleep in People With Epilepsy
Brief Title: Sleep and Rehearsal-Driven Memory in Epilepsy
Acronym: CORESOM-EPI
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_0188; 2025-A00510-49 (Other: ID-RCB)
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Epilepsy; Memory Consolidation
Keywords: Epilepsy; Memory consolidation; Sleep; Reharsal; Reactivation
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- WAKE - SLEEP: This group will start with the condition 1 " wake " (encoding+immediate recall in the morning (8 :00am) and delayed recall in the evening (8 :00pm)) and will end with the condition 2 " sleep " : (encoding+immediate recall in the evening (8 :00pm) and delayed recall in the morning (8 :00am))
  Interventions: Other: Cognitive memory task on a computer; Other: Eye tracking; Other: Questionnaires on task-related fatigue; Other: Questionnaire on task difficulty; Other: Karolinska scale
- SLEEP-WAKE: This group will start with the condition 2 " sleep "and will end with the condition 1 " wake "
  Interventions: Other: Cognitive memory task on a computer; Other: Eye tracking; Other: Questionnaires on task-related fatigue; Other: Questionnaire on task difficulty; Other: Karolinska scale

INTERVENTIONS:
Other: Cognitive memory task on a computer — Encoding: (1) Participants will learn 60 associations between pairs of items (cue and target) that are presented sequentially at unique locations on a screen, in a given context. 30 pairs are presented once, and 30 pairs are presented repeatedly (4 times).
  (2) After learning, the first recall phase begins after a short delay of 30 minutes: 50% of the pairs are tested in a similar way, this time with an assessment of contextual memory.
  (3) The remaining 50% of pairs are tested after a 12-hour delay, involving either a day awake (condition 1) or a night asleep (condition 2).
Other: Eye tracking — Eye-tracking will be carried out during the task to ensure that participants are focused on the task (quantification of the number and duration of eye fixations in the area of interest corresponding to the target presentation)
Other: Questionnaires on task-related fatigue — Questionnaire on task-related fatigue (Likert-scale) will be completed by participants between blocks of items during the task
Other: Questionnaire on task difficulty — Questionnaires on task difficulty (Likert-scale) will be completed by participants at the end of the task
Other: Karolinska scale — Participants' state of sleepiness will be assessed at the beginning of each stage (encoding, immediate recall, delayed recall) using the Karolinska sleepiness scale

SUMMARY:
Memory consolidation transforms unstable memory traces into lasting representations, a process enhanced by both sleep and rehearsal during learning. Rehearsal is thought to accelerate consolidation by inducing memory reactivations that resemble those occurring during sleep. However, the respective mechanisms of sleep- and rehearsal-induced consolidation-and their potential interactions-remain poorly understood, especially in patients with temporal lobe epilepsy, where rehearsal might help compensate for memory deficits linked to hippocampal dysfunction, and where sleep may exacerbate epileptic activity. The CORESOM-EPI study aims to compare the effects of rehearsal and sleep on memory consolidation in patients undergoing video-EEG monitoring. Participants will learn "object-place" associations under two conditions (single versus repeated encoding), with memory tested immediately and again after a 12-hour delay. This delay will either include a full day awake or a night of sleep, allowing direct comparison of sleep- and rehearsal-related consolidation effects. Each participant will perform the task twice, with "wake" and "sleep" condition, in a balanced order. As a preliminary phase of the CRIMES study (ANR-DFG 2024), CORESOM-EPI will help assess how sleep and rehearsal influence memory consolidation in epilepsy. It will also serve to adapt the behavioral task for clinical use, paving the way for a future intracranial EEG investigations that will explore the neural networks involved and their modulation by epileptic activity.

ELIGIBILITY:
Inclusion Criteria:

* Patient with epilepsy (any type of epilepsy)
* Hospitalized for video-EEG recording lasting at least 4 days
* Aged 18-65 years

Exclusion Criteria:

* Major cognitive impairment other than memory deficit
* Refusal to participate
* Pregnant women, women in labor or nursing mothers
* Persons deprived of their liberty by judicial or administrative decision
* Persons under psychiatric care
* Persons admitted to a health or social institution for purposes other than research
* Adults under legal protection (guardianship, curatorship)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with epilepsy admitted to the Functional Neurology and Epileptology Department of the Hospices Civils de Lyon (University Hospital) for video-EEG monitoring will be invited by the investigating physician to participate in the study. If patients wish to take part, they will be asked to perform a cognitive task.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in the percentage of object categories recalled (vs. not recalled) between immediate (30 min after learning) and delayed (12h after learning) recall for rehearsed versus non-rehearsed items. | Day 2
  The impact of rehearsal on object category recognition in an object-place learning paradigm is assessed.
  For the primary outcome, data from the 2 conditions ("wake" and "sleep" during the 12h period between immediate and delayed recall) will be pooled. Each participant will take part in the wake and sleep condition over 4 days (2 conditions separated by at least 24h), in a balanced order between participants.
Change in the percentage of object categories recalled (vs. not recalled) between immediate (30 min after learning) and delayed (12h after learning) recall for rehearsed versus non-rehearsed items. | Day 2 + 12 hours
  The impact of rehearsal on object category recognition in an object-place learning paradigm is assessed.
  For the primary outcome, data from the 2 conditions ("wake" and "sleep" during the 12h period between immediate and delayed recall) will be pooled. Each participant will take part in the wake and sleep condition over 4 days (2 conditions separated by at least 24h), in a balanced order between participants.
Change in the percentage of object categories recalled (vs. not recalled) between immediate (30 min after learning) and delayed (12h after learning) recall for rehearsed versus non-rehearsed items. | Day 2 + 36 hours
  The impact of rehearsal on object category recognition in an object-place learning paradigm is assessed.
  For the primary outcome, data from the 2 conditions ("wake" and "sleep" during the 12h period between immediate and delayed recall) will be pooled. Each participant will take part in the wake and sleep condition over 4 days (2 conditions separated by at least 24h), in a balanced order between participants.
Change in the percentage of object categories recalled (vs. not recalled) between immediate (30 min after learning) and delayed (12h after learning) recall for rehearsed versus non-rehearsed items. | Day 2 + 48 hours
  The impact of rehearsal on object category recognition in an object-place learning paradigm is assessed.
  For the primary outcome, data from the 2 conditions ("wake" and "sleep" during the 12h period between immediate and delayed recall) will be pooled. Each participant will take part in the wake and sleep condition over 4 days (2 conditions separated by at least 24h), in a balanced order between participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de neurologie fonctionnelle et d'épileptologie, Hôpital neurologique Pierre Wertheimer, Bron, France